CLINICAL TRIAL: NCT06396117
Title: Relationship Between Anogenital Distance and Serum AMH and mTESE Associated With or Without Klinefelter Syndrome
Brief Title: Relationship Between Anogenital Distance, Serum AMH, and mTESE in Klinefelter Syndrome
Acronym: KS
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Wael Ragab, Lecturer, Cairo University
Other Study IDs: AND AMH
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Azoospermia Anogenital Distance AMH

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients who have KS: Group one is patients with Klinefelter syndrome confirmed as 47, XXY on karyotyping undergoing mTESE for non-obstructive azoospermia
  Interventions: Other: mTESE (microscopic testicular sperm extraction)
- Patient who does not have KS: Group two consists of patients with a normal karyotyping undergoing mTESE for non-obstructive azoospermia
  Interventions: Other: mTESE (microscopic testicular sperm extraction)

INTERVENTIONS:
Other: mTESE (microscopic testicular sperm extraction) — Microdissection Testicular Sperm Extraction (mTESE) is a surgical procedure used to retrieve sperm from the testicles of men with non-obstructive azoospermia (NOA). It involves:
  1. Testicular biopsy: Removing a small sample of testicular tissue.
  2. Microscopic examination: Examining the tissue under a microscope to identify areas with sperm production.
  3. Sperm extraction: Dissecting out individual sperm cells from the testicular tissue.
  This technique allows for:
  * More accurate identification of sperm-containing areas
  * Lower risk of damage to surrounding testicular tissue
  * Potential for higher sperm retrieval rates compared to conventional method

SUMMARY:
Azoospermia, the absence of sperm in the ejaculate, affects approximately 1% of males and 15% of infertile men. Non-obstructive azoospermia (NOA) accounts for 60% of azoospermic patients, who rely solely on testicular sperm extraction (TESE) surgery for sperm harvesting. While conventional TESE (cTESE) and microdissection TESE (mTESE) are preferred methods, the lack of predictive biomarkers for successful sperm retrieval (SR) renders treatment unnecessary for many NOA males. However, research suggests that anti-Mullerian hormone (AMH) and anogenital distance (AGD) may serve as predictors of positive SR at mTESE in NOA males. AGD, a marker of fetal androgen disruption and adult outcomes, may also assess male reproductive potential by predicting normal genital growth and sperm creation. A cross-sectional study found a positive correlation between AGD and total sperm count, concentration, and motility in infertile men aged 25-38, providing valuable prognostic insights for azoospermic men.

DETAILED DESCRIPTION:
Azoospermia, which is defined as the lack of spermatozoa in the ejaculate, is a condition that affects around one percent of males and fifteen percent of men who are infertile. Sixty percent of azoospermic patients are affected by non-obstructive azoospermia, often known as NOA.

To harvest sperm for assisted reproductive technology (ART), this subset of men has no other choice except to undergo testicular sperm extraction (TESE) surgery.

Conventional TESE (cTESE) and microdissection TESE (mTESE) are the most preferred procedures in terms of sperm retrieval (SR) rates and the decrease of damage caused by excision. Studies have revealed varying percentages of positive SR, ranging from thirty percent to sixty percent.

This treatment is not necessary for a significant number of NOA boys because there are no biomarkers or procedures that are clinically acceptable that can predict a positive SR score at mTESE.

According to earlier research, anti-mullerian hormone (AMH), which is a homodimeric glycoprotein belonging to the family of transforming growth factor-b, has the potential to predict either a positive or negative significant difference (SR) at mTESE in iNOA. Throughout the course of development, Sertoli cells (SCs) secrete Amyloid-beta (AMH) in order to regress the Mullerian ducts and ensure that male sex differentiation occurs. AMH levels drop significantly when the development of puberty in males and the maturation of SCs occurs. It has been suggested that this hormone, which is solely produced by spermatocytes in males, can be used as an indirect marker of spermatogenesis, maturation of spermatocytes, and immaturity of the prepubertal testes.

A noninvasive method known as anogenital distance has recently been applied for the purpose of predicting and diagnosing disorders. There are two different measurements of the anogenital distance (AGD) for both men and women. AGD is a marker that indicates fetal androgen dysregulation as well as negative effects in adulthood. AGD is a unique method that can be used to evaluate the reproductive potential of males because it has the capacity to predict normal male genital growth and the production of sperm. It may also assist medical professionals in providing prognostic information to men who are azoospermic.

AGD AS was found to have a positive correlation with total sperm count, concentration, and motility in a cross-sectional study where the participants were infertile men between the ages of 25 and 38.

ELIGIBILITY:
Inclusion Criteria:

* All NOA patients underwent mTESE at the Andrology department, Kasr Al-Ainy hospitals

Exclusion Criteria:

* patients with

  1. Obstructive azoospermia
  2. Retrograde Ejaculation
  3. Men with hypogonadotropic hypogonadism

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Male patients with non-obstructive azoospermia of any age group suffering from infertility who did two successive semen analyses at least two weeks apart showing no sperms in ejaculate with normal or elevated gonadotrophic hormones and will undergo Testicular Sperm Extraction operation at Andrology Department, Kasr Al Ainy hospital Cairo University.
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Relation of AGD of males with azoospermia (with or without KS) to mTESE outcome | 1 months
  Higher AGD might be correlated to higher sperm retrieval
Relation of AMH in males with azoospermia (with or without KS) to mTESE outcome | 1 month
  Higher AMH might be correlated to higher sperm retrieval

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy, Cairo, Please Select A Region, State Or Province., Egypt

IPD SHARING:
Plan to Share IPD: No